Study Protocol of a Randomized Controlled Trial of an Online Self-care Training Program to Reduce Burnout and Promote Work Engagement in Chilean Psychologists: MAGO Study

NCT04462484

September 29th, 2020.

## DATA PROTECTION

- Data controller: University of Padova.
- Organizational referent for privacy: Dr. Sabrina Cipolletta.
- UNIPD people authorized to process the data: Pablo Hernández Lillo, Dr. Caterina Novara.
- Data processor: Dr. Felipe Gálvez Sánchez (University of Chile), Isabel Wolnitzky (University of Chile).





## INFORMED CONSENT (English version)

Study protocol of a randomized controlled trial of an online self-care training program to reduce burnout and promote work engagement in Chilean psychologists: MAGO Study

## I. INFORMATION

You have been invited to participate in the research "Study protocol of a randomized controlled trial of an online self-care training program to reduce burnout and promote work engagement in Chilean psychologists: MAGO Study". The objective of the study is to determine the Efficacy of the intervention Online Guided Self-Care Model (MAGO). This activity corresponds to an individual occupational intervention directed by videoconference, which lasts six sessions on a weekly basis. By promoting self-care behaviors, it is expected to reduce the levels of burnout at work and increase work commitment in clinical psychologists working in Chile. You have been invited because you are currently working as a clinical psychologist in the public sector.

The researcher responsible for this study is Pablo Cristóbal Hernández Lillo, a student of the Brain, Mind and Computer Science PhD program at the University of Padua, Italy. The research is sponsored by the Conicyt Doctoral Scholarship.

In deciding to participate in this research, it is important that you consider the following information. Feel free to ask any matter that is unclear to you:

Participation: Participants will be randomly assigned to a control group and an intervention group.

If you are assigned to the intervention group, you will be invited to participate in six sessions of 45 minutes (on a weekly basis) of videoconference where you will discuss the aspects of self-care and how to incorporate them into your own work as a clinical psychologist. There will be some optional tasks between sessions such as activity planning or journal writing. Video conference hours will be agreed and scheduled in advance by email. Sessions can be interrupted and resumed in coordination with the researcher.

All participants (assigned to control and intervention groups) will receive online questionnaires three times: two weeks before the intervention, two weeks after the intervention, and six months after the intervention. The questionnaires are as follows:

BAI Anxiety
 BDI-IA Depression
 MBI-HSS Burnout syn

MBI-HSS Burnout symptoms
 UWES-17 Work engagement
 SCAP Self-care behaviors
 GHQ-12 General health

7. MSPSS Perceived social support

**Risks**: Your participation does not entail risks for you.

**Benefits**: You will not receive any direct benefits or rewards for participating in this study. However, your participation will allow you to generate information to know indicators of your relationship with work and some related aspects of your mental health.





If you are assigned to the intervention group, you may benefit from incorporating self-care behaviors into your own work context.

If you were not assigned to the intervention group and the final results indicate that the proposed activity is effective, we promise to contact you to offer to participate in the intervention (videoconference sessions). If you decide to participate, all the videoconference sessions of the intervention will be given to you free of charge.

**Voluntariness**: Your participation is absolutely voluntary. You are free to answer the questions you want, as well as to stop participating at any time you want. This will not be detrimental to you.

**Confidentiality**: All your opinions will be confidential, and kept strictly confidential. Your personal information and results will be kept confidential and stored separately. For this, a code will be assigned to each participant and only researchers will have access to the data. In the presentations and publications of this research, your name will not appear associated with any particular opinion.

The videoconference sessions will be supported in audio and video, and can only be reviewed by researchers. These files will be deleted once the study is completed. Therefore, the videos will not be used in results or publications.

**Knowledge of the results**: You have the right to know the results of this investigation, which will be sent to your email. For this reason, we ask you to provide us with a contact email at the end of this document.

**Contact information**: If you require more information, or communicate for any reason related to this research, you can contact the Investigator Responsible for this study

Pablo Hernandez

Email: p.hernandezlillo@gmail.com

You can also contact the Responsible Investigator located in Chile:

Prof. Felipe Gálvez Sánchez
Academic Department of Psychology
University of Chile
Phone: (56-2) 9787806
Email: galvezsanghez@ughilo.gl

Email: galvezsanchez@uchile.cl

Address

1045 Ignacio Carrera Pinto Avenue, Ñuñoa, Santiago, Chile.

You can also contact the Chairman of the Research Ethics Committee that approved this study:

Prof. Dr. Uwe Kramp Denegri

President

Research Ethics Committee Faculty of Social Sciences

University of Chile

Phone: (56-2) 29772443

Address: Av. Ignacio Carrera Pinto 1045, Ñuñoa, Santiago. Faculty of Social Sciences, Building A,

Deanship Department. University of Chile.

Email: comite.etica@facso.cl



COMITÉ DE ETICA DE LA INVESTIGACIÓN Facultad de Ciencias Sociales UNIVERSIDAD DE CHILE

## **II. INFORMED CONSENT FORM**

| I,, a protocol of a randomized controlled trial of an online se and promote work engagement in Chilean psychologis here. | elf-care training program to reduce burnout |
|---|---|
| I declare that I have read (or had read to me) and (have participation in this study. I have had the opportur been answered. I have no doubts about it. | |
| I agree to participate in online questionnaires: Yes | No |
| I agree to participate in videoconference sessions: Yes | SNo |
| Participant signature Res | ponsible Investigator signature |
| Place and date: | |
| Email for the return of the information: | |
| This document consists of four pages and is signed in | two copies, leaving one copy in each part. |